CLINICAL TRIAL: NCT05255692
Title: Pilot Study: Apllicability of an fMRI Protocol for Incontinence Research
Brief Title: Brain Activity During Bladder Filling: Pilot Study of an fMRI Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BC-10572
Record Dates: First submitted 2022-01-24; First posted 2022-02-24 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: fMRI Research
Keywords: Bladder control; functional magnetic resonance imaging
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complete evaluation UDO and fMRI (Experimental): Evaluation including both urodynamic evaluation and functional MRI testing
  Interventions: Diagnostic Test: invasive urodynamic evaluation; Diagnostic Test: functional magnetic resonance imaging during bladder filling

INTERVENTIONS:
Diagnostic Test: invasive urodynamic evaluation — Invasive urodynamic evaluation to define maximum cystometric capacity. By means of catheterisation the bladder gets filled and volumes en pressures are measured.
  Other Names: UDO
Diagnostic Test: functional magnetic resonance imaging during bladder filling — Functional MRI is used to capture brain activity during tasks. The task in the current study is bladder infusion and withdrawal by means of the INFSYS-2 infusion/withdrawal pump (Leitner et al. 2017)
  Other Names: fMRI

SUMMARY:
Urinary incontinence is the most frequently observed lower urinary tract symptom (LUTS) in children with cerebral palsy (CP) (Samijn et al., 2016).

Higher brain centers responsible for bladder function may be related to the presence of incontinence.

The current pilot study is the first study of a research project focusing on correlations between brain damage and incontinence.

DETAILED DESCRIPTION:
Urinary incontinence is the most frequently observed lower urinary tract symptom (LUTS) in children with cerebral palsy (CP) (Samijn et al., 2016). Being more or completely dry could improve the quality of life and health status of the child and the social environment.

Higher brain centers responsible for bladder function may be related to the presence of incontinence. These higher brain centers could be correlated to the brain damage seen in children with CP.

The current pilot study is the first study of a research project focusing on correlations between brain damage and incontinence. The study wants to validate if the defined fMRI paradigm can provide correct information concerning brain activity during bladder filling, to ensure usable results and comply with ethical demands for testing in children, the protocol will be tested and results validated during the pilot study with healthy adults. During the fMRI study, the bladder will be filled until FSF and NDV. Functional MRI-data will be obtained during the filling and emptying phase of the bladder on both volumes

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* lower or upper urinary tract dysfunction

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Activated brain regions demonstrating brain activity | through study completion, an average of 6 weeks
  fMRI brain imaging data will be analyzed using FMRIB Software Library v6.0 (FSL).

CONTACTS AND LOCATIONS:
Overall Officials: Bieke Samijn, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No